CLINICAL TRIAL: NCT07274982
Title: The Importance of Modified EASIX Score in Determining Severity of Erectile Dysfunction - A Single-Center Retrospective Case-Control Study
Brief Title: The Predictive Value of Modified EASIX Score for Determining Erectile Dysfunction Severity
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Collaborators: Ministry of Health, Turkey (Other Government)
Responsible Party: Principal Investigator, okkes zortuk, Principal Investigator, Ataturk University
Other Study IDs: ZTKLAB03112025KUGOEK2520UROLGY
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Erectile Dysfunctions; Endothelial Dysfunction; Inflammation
Keywords: Erectile Dysfunctions; EASIX; modified EASIX; IIEF-5; endothelial inflammation
MeSH Terms: conditions — Erectile Dysfunction; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erectile Dysfunction Group: Erectile Dysfunction Group
  Interventions: Other: IIEF-5; Other: mEASIX
- Non-Erectile Dysfunction Group: Non-Erectile Dysfunction Group
  Interventions: Other: IIEF-5; Other: mEASIX

INTERVENTIONS:
Other: IIEF-5 — IIEF-5: The erectile dysfunction status of patients will be analyzed with the International Index of Erectile Function-5.
Other: mEASIX — Endothelial function will be evaluated with mEAX.

SUMMARY:
This retrospective single-center case-control study evaluates whether the Modified EASIX score (LDH × CRP / Platelets), calculated from routine blood tests, predicts severity of erectile dysfunction (ED) as measured by the IIEF-5 questionnaire. Medical records from January 1, 2024 to September 30, 2025 will be reviewed. Patients will be classified by IIEF-5 (≤21 = ED; ≥22 = no ED) and Modified EASIX distributions and predictive performance (ROC/AUC) will be compared between groups. No additional interventions will be performed.

DETAILED DESCRIPTION:
This retrospective observational study will include adult male patients aged 18-65 attending the urology outpatient clinic. Demographic data, comorbidities, IIEF-5 scores and routine laboratory results (LDH, CRP, platelet count and other routine biochemistry/hematology) obtained during routine follow-up will be extracted from medical records covering January 2024-September 2025. The Modified EASIX score will be computed as: LDH × CRP / Platelets. Patients will be grouped according to IIEF-5: ED group (IIEF-5 ≤21) and non-ED group (IIEF-5 ≥22). Primary analyses include group comparisons of Modified EASIX, correlation analyses with IIEF-5, logistic regression for association and ROC analysis to evaluate discriminatory performance and optimal cut-offs. Analyses will use IBM SPSS 27 and GraphPad Prism 9. No changes to patient management were made for study purposes; no additional sampling or interventions were performed.

ELIGIBILITY:
Inclusion Criteria:

Male patients aged 18-65. Followed at the urology outpatient clinic with a documented IIEF-5 questionnaire.

Available routine laboratory data including LDH, CRP and platelet count within the study period (Jan 1, 2024 - Sep 30, 2025).

Exclusion Criteria:

Use of penile prosthesis. Patients without an organic ED diagnosis when relevant (per protocol: "Patients without an organic ED diagnosis will be excluded from the study").

Missing essential data for Modified EASIX calculation or IIEF-5.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only self-identified male participants aged 18-65 are eligible, as the study focuses on erectile dysfunction, a condition specific to individuals with male genital anatomy.
Study Population: Adult male patients aged 18-65 who attended the urology outpatient clinic and had documented IIEF-5 scores and routine laboratory results (LDH, CRP, platelet count) between January 2024 and September 2025. The study includes both patients with erectile dysfunction (IIEF-5 ≤ 21) and those without erectile dysfunction (IIEF-5 ≥ 22), using retrospectively collected medical records from a single center (Defne State Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Difference in Modified EASIX score between ED and non-ED groups | Retrospective records from Jan 1, 2024 to Sep 30, 2025.
  Mean Modified EASIX (LDH × CRP / Platelets) in each group. Group comparison (t-test) and effect size.
Difference in Modified EASIX score between ED and non-ED groups | Time Frame: Retrospective records from Jan 1, 2024 to Sep 30, 2025.
  Median Modified EASIX (LDH × CRP / Platelets) in each group. Group comparison (Mann-Whitney U) and effect size.

CONTACTS AND LOCATIONS:
Locations (1):
- Defne State Hospital, Hatay, Defne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared because the study is based on retrospective medical records containing sensitive personal health information. Due to privacy concerns and institutional data-protection regulations, de-identified datasets cannot be released outside the research team.

REFERENCES:
- [Result] Zinczuk A, Rorat M, Simon K, Jurek T. EASIX, Modified EASIX and Simplified EASIX as an Early Predictor for Intensive Care Unit Admission and Mortality in Severe COVID-19 Patients. J Pers Med. 2022 Jun 21;12(7):1022. doi: 10.3390/jpm12071022. PMID 35887519
- [Result] Pennisi M, Sanchez-Escamilla M, Flynn JR, Shouval R, Alarcon Tomas A, Silverberg ML, Batlevi C, Brentjens RJ, Dahi PB, Devlin SM, Diamonte C, Giralt S, Halton EF, Jain T, Maloy M, Mead E, Palomba ML, Ruiz J, Santomasso B, Sauter CS, Scordo M, Shah GL, Park JH, Yanez San Segundo L, Perales MA. Modified EASIX predicts severe cytokine release syndrome and neurotoxicity after chimeric antigen receptor T cells. Blood Adv. 2021 Sep 14;5(17):3397-3406. doi: 10.1182/bloodadvances.2020003885. PMID 34432870